CLINICAL TRIAL: NCT04187144
Title: A Phase III, Randomized, Multicenter, Parallel-Group, Double-Blind, Double-Dummy Study in Adolescent and Adult Female Participants Comparing the Efficacy and Safety of Gepotidacin to Nitrofurantoin in the Treatment of Uncomplicated Urinary Tract Infection (Acute Cystitis)
Brief Title: Comparative Study to Evaluate Efficacy and Safety of Gepotidacin to Nitrofurantoin in Treatment of Uncomplicated Urinary Tract Infection (UTI)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 212390; 2020-000553-27 (EudraCT Number)
Record Dates: First submitted 2019-12-03; First posted 2019-12-05 (Actual); Results first posted 2023-07-18 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Urinary Tract Infections
Keywords: Acute cystitis; Efficacy; Gepotidacin; Nitrofurantoin; Urinary Tract Infection; Simple cystitis
MeSH Terms: conditions — Urinary Tract Infections | interventions — gepotidacin; Nitrofurantoin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Gepotidacin (Experimental): Participants will be administered oral doses of 1500 milligrams (mg) gepotidacin plus nitrofurantoin matching placebo BID; approximately every 12 hours for 5 days.
  Interventions: Drug: Gepotidacin; Drug: Placebo matching nitrofurantoin
- Nitrofurantoin (Active Comparator): Participants will be administered oral doses of 100 mg nitrofurantoin plus gepotidacin matching placebo BID; approximately every 12 hours for 5 days.
  Interventions: Drug: Nitrofurantoin; Drug: Placebo matching gepotidacin

INTERVENTIONS:
Drug: Gepotidacin — Gepotidacin will be available as tablets at a unit dose strength of 750mg. Participants will administer two 750 mg tablets, BID. Each dose will be taken with water after consumption of food.
  Arms: Gepotidacin
Drug: Placebo matching nitrofurantoin — Placebo matching nitrofurantoin will be available as over-encapsulated unit-dose capsules. Participants will administer 1 capsule BID. Each dose should be taken with water after consumption of food.
  Arms: Gepotidacin
Drug: Nitrofurantoin — Nitrofurantoin will be available as over-encapsulated 100 mg capsules containing 25 mg nitrofurantoin macrocrystals and 75 mg nitrofurantoin. Participants will administer one 100 mg capsule, BID. Each dose should be taken with water after consumption of food.
  Arms: Nitrofurantoin
Drug: Placebo matching gepotidacin — Placebo matching gepotidacin will be available as unit-dose gepotidacin placebo-to-match tablet. Participants will administer two tablets, BID. Each dose should be taken with water after consumption of food.
  Arms: Nitrofurantoin

SUMMARY:
The study will be conducted to evaluate the therapeutic response (combined per participant microbiological and clinical response) of oral gepotidacin compared to oral nitrofurantoin for treatment of uncomplicated UTI (acute cystitis) in adolescent and adult female participants.

ELIGIBILITY:
Inclusion Criteria:

* The participant is >=12 years of age at the time of signing the informed consent/assent and has a body weight >=40 kilogram (kg).
* The participant has 2 or more of the following clinical signs and symptoms of acute cystitis with onset <96 hours prior to study entry: dysuria, frequency, urgency, or lower abdominal pain.
* The participant has nitrite or pyuria (greater than [>]15 white blood cell [WBC]/high-power field [HPF]) or the presence of 3 plus (+)/large leukocyte esterase) from a pretreatment clean-catch midstream urine sample based on local laboratory procedures.
* The participant is female.
* The participant is capable of giving signed informed consent/assent.

Exclusion Criteria:

* The participant resides in a nursing home or dependent care type-facility.
* The participant has a body mass index >=40.0 kilogram per meter square (kg/m^2) or a body mass index >=35.0 kg/m^2 and is experiencing obesity-related health conditions such as uncontrolled high blood pressure or uncontrolled diabetes.
* The participant has a history of sensitivity to the study treatment, or components thereof, or a history of a drug or other allergy that, in the opinion of the investigator or medical monitor, contraindicates her participation.
* The participant is immunocompromised or has altered immune defenses that may predispose the participant to a higher risk of treatment failure and/or complications.
* The participant has any of the following:

  1. Poorly controlled asthma or chronic obstructive pulmonary disease; Acute severe pain,; Active peptic ulcer disease; Parkinson disease; Myasthenia gravis; Or
  2. Known acute porphyria.
  3. Any surgical or medical condition (active or chronic) that may interfere with drug absorption, distribution, metabolism, or excretion of the study intervention .
* The participant has a known glucose-6 phosphate dehydrogenase deficiency.
* The participant has a serious underlying disease that could be imminently life threatening, or the participant is unlikely to survive for the duration of the study period.
* The participant has acute cystitis that is known or suspected to be due to fungal, parasitic, or viral pathogens; or known or suspected to be due to Pseudomonas aeruginosa or Enterobacterales (other than Escherichia coli) as the contributing pathogen.
* The participant has symptoms known or suspected to be caused by another disease process, such as asymptomatic bacteriuria, overactive bladder, chronic incontinence, or chronic interstitial cystitis, that may interfere with the clinical efficacy assessments or preclude complete resolution of acute cystitis symptoms.
* The participant has an anatomical or physiological anomaly that predisposes the participant to UTIs or may be a source of persistent bacterial colonization, including calculi, obstruction or stricture of the urinary tract, primary renal disease (for example [e.g.], polycystic renal disease), or neurogenic bladder, or the participant has a history of anatomical or functional abnormalities of the urinary tract (e.g., chronic vesico-ureteral reflux, detrusor insufficiency).
* The participant has an indwelling catheter, nephrostomy, ureter stent, or other foreign material in the urinary tract.
* The participant who, in the opinion of the investigator, has an otherwise complicated UTI, an active upper UTI (e.g., pyelonephritis, urosepsis), signs and symptom onset >=96 hours before study entry, or a temperature >=101.4 degree Fahrenheit (>=38 Degrees Celsius [C]), flank pain, chills, or any other manifestations suggestive of upper UTI.
* The participant has known anuria, oliguria, or significant impairment of renal function (creatinine clearance <60 milliliters per minute (mL/min) or clinically significant elevated serum creatinine as determined by the investigator).
* The participant presents with vaginal discharge at Baseline (e.g., suspected sexually transmitted disease).
* The participant has congenital long QT syndrome or known prolongation of the QTc interval.
* The participant has uncompensated heart failure.
* The participant has severe left ventricular hypertrophy.
* The participant has a family history of QT prolongation or sudden death.
* The participant has a recent history of vasovagal syncope or episodes of symptomatic bradycardia or brady arrhythmia within the last 12 months.
* The participant is taking QT-prolonging drugs or drugs known to increase the risk of torsades de pointes (TdP) per the www.crediblemeds.org. "Known Risk of TdP" category at the time of her Baseline Visit, which cannot be safely discontinued from the Baseline Visit to the TOC Visit; or the participant is taking a strong cytochrome P450 enzyme 3A4 (CYP3A4) inhibitor.
* For any participant >=12 to <18 years of age, the participant has an abnormal ECG reading.
* The participant has a QTc >450 msec or a QTc >480 msec for participants with bundle-branch block.
* The participant has a documented or recent history of uncorrected hypokalemia within the past 3 months.
* The participant has a known ALT value >2 times upper limit of normal (ULN).
* The participant has a known bilirubin value >1.5 times ULN (isolated bilirubin >1.5 times ULN is acceptable if bilirubin is fractionated and direct bilirubin <35 percent [%]).
* The participant has cirrhosis or current unstable liver or biliary disease per investigator assessment defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, or persistent jaundice.
* The participant has a previous history of cholestatic jaundice/hepatic dysfunction associated with nitrofurantoin.
* The participant has received treatment with other systemic antimicrobials or systemic antifungals within 1 week before study entry.

Min Age: 12 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 1606 (Actual)
Dates: Start 2020-04-23 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (102):
- United States (69):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Homewood, Alabama
  - GSK Investigational Site, Huntsville, Alabama
  - GSK Investigational Site, Gilbert, Arizona
  - GSK Investigational Site, Peoria, Arizona
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, La Mesa, California
  - GSK Investigational Site, Modesto, California
  - GSK Investigational Site, Northridge, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, Valencia, California
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Apollo Beach, Florida
  - GSK Investigational Site, Boynton Beach, Florida
  - GSK Investigational Site, Clearwater, Florida
  - GSK Investigational Site, Coconut Creek, Florida
  - GSK Investigational Site, Gainesville, Florida
  - GSK Investigational Site, Hialeah, Florida
  - GSK Investigational Site, Lake Worth, Florida
  - GSK Investigational Site, Leesburg, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Ormond Beach, Florida
  - GSK Investigational Site, Palm Springs, Florida
  - GSK Investigational Site, Pembroke Pines, Florida
  - GSK Investigational Site, Plant City, Florida
  - GSK Investigational Site, Sweetwater, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Blackfoot, Idaho
  - GSK Investigational Site, Boise, Idaho
  - GSK Investigational Site, Meridian, Idaho
  - GSK Investigational Site, Hanover, Maryland
  - GSK Investigational Site, Fall River, Massachusetts
  - GSK Investigational Site, Butte, Montana
  - GSK Investigational Site, Lincoln, Nebraska
  - GSK Investigational Site, East Orange, New Jersey
  - GSK Investigational Site, Lawrenceville, New Jersey
  - GSK Investigational Site, Mount Laurel, New Jersey
  - GSK Investigational Site, Brooklyn, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Cary, North Carolina
  - GSK Investigational Site, Wilmington, North Carolina
  - GSK Investigational Site, Winston-Salem, North Carolina
  - GSK Investigational Site, Fargo, North Dakota
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Dayton, Ohio
  - GSK Investigational Site, Eugene, Oregon
  - GSK Investigational Site, Bala-Cynwyd, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Lancaster, South Carolina
  - GSK Investigational Site, Union, South Carolina
  - GSK Investigational Site, Milan, Tennessee
  - GSK Investigational Site, New Tazewell, Tennessee
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Katy, Texas
  - GSK Investigational Site, Mesquite, Texas
  - GSK Investigational Site, Missouri City, Texas
  - GSK Investigational Site, North Richland Hills, Texas
  - GSK Investigational Site, Plano, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Bountiful, Utah
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, St. George, Utah
  - GSK Investigational Site, Richmond, Virginia
- Australia (3):
  - GSK Investigational Site, Maroubra, New South Wales
  - GSK Investigational Site, Sydney, New South Wales
  - GSK Investigational Site, Tarragindi, Queensland
- Bulgaria (10):
  - GSK Investigational Site, Gabrovo
  - GSK Investigational Site, Haskovo
  - GSK Investigational Site, Kyustendil
  - GSK Investigational Site, Montana
  - GSK Investigational Site, Pleven
  - GSK Investigational Site, Rousse
  - GSK Investigational Site, Shumen
  - GSK Investigational Site, Sofia
  - GSK Investigational Site, Stara Zagora
  - GSK Investigational Site, Targovisthe
- India (10):
  - GSK Investigational Site, Aurangabad
  - GSK Investigational Site, Chandrapur
  - GSK Investigational Site, Hyderabad
  - GSK Investigational Site, Mumbai
  - GSK Investigational Site, Nagpur
  - GSK Investigational Site, Nashik
  - GSK Investigational Site, New Delhi
  - GSK Investigational Site, Pune
  - GSK Investigational Site, Rajkot
  - GSK Investigational Site, Surat
- Poland (4):
  - GSK Investigational Site, Katowice
  - GSK Investigational Site, Ostrowiec Świętokrzyski
  - GSK Investigational Site, Świdnik
  - GSK Investigational Site, Warsaw
- South Korea (6):
  - GSK Investigational Site, Ansan-si
  - GSK Investigational Site, Goyang-si, Gyeonggi-do
  - GSK Investigational Site, Hwasun-gun, Jeollanam-do
  - GSK Investigational Site, Incheon
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Suwon

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Wagenlehner F, Kaye KS, Talan DA, Sheets AJ, Scangarella-Oman NE, Jarvis E, Dennison J, Janmohamed S, Helgeson M, Perry C. Impact of updated regulatory guidelines on study results in contemporary uncomplicated urinary tract infection clinical trials and implications for trial conduct and drug development: a comparative analysis with EAGLE-2 and EAGLE-3. Contemp Clin Trials Commun. 2025 Nov 18;48:101572. doi: 10.1016/j.conctc.2025.101572. eCollection 2025 Dec. PMID 41399629
- [Derived] Scangarella-Oman NE, Butler DL, Breton J, Brown D, Kasapidis C, Sheets AJ. Efficacy and in vitro activity of gepotidacin against bacterial uropathogens, including subsets with molecularly characterized resistance mechanisms and genotypes/epidemiological clones, in females with uncomplicated urinary tract infections: results from two global, pivotal, phase 3 trials (EAGLE-2 and EAGLE-3). Antimicrob Agents Chemother. 2025 Oct;69(10):e0163924. doi: 10.1128/aac.01639-24. Epub 2025 Sep 9. PMID 40924012
- [Derived] Scangarella-Oman NE, Butler DL, Breton J, Brown D, Kasapidis C, Millns H, Huang C, Perry CR, Sheets AJ, Dennison J, Janmohamed S. Efficacy and in vitro activity of gepotidacin against bacterial uropathogens, including drug-resistant phenotypes, in females with uncomplicated urinary tract infections: results from two global, pivotal, phase 3 trials (EAGLE-2 and EAGLE-3). Antimicrob Agents Chemother. 2025 Oct;69(10):e0164024. doi: 10.1128/aac.01640-24. Epub 2025 Sep 9. PMID 40924001
- [Derived] Hackel MA, Karlowsky JA, Sahm DF, West JM, Scangarella-Oman NE. In vitro activity of gepotidacin against urinary tract infection isolates of Enterobacterales, Enterococcus faecalis, and Staphylococcus saprophyticus. Antimicrob Agents Chemother. 2025 Jun 4;69(6):e0029625. doi: 10.1128/aac.00296-25. Epub 2025 May 15. PMID 40372095
- [Derived] Wagenlehner F, Perry CR, Hooton TM, Scangarella-Oman NE, Millns H, Powell M, Jarvis E, Dennison J, Sheets A, Butler D, Breton J, Janmohamed S. Oral gepotidacin versus nitrofurantoin in patients with uncomplicated urinary tract infection (EAGLE-2 and EAGLE-3): two randomised, controlled, double-blind, double-dummy, phase 3, non-inferiority trials. Lancet. 2024 Feb 24;403(10428):741-755. doi: 10.1016/S0140-6736(23)02196-7. Epub 2024 Feb 8. PMID 38342126
- [Derived] Perry C, Hossain M, Powell M, Raychaudhuri A, Scangarella-Oman N, Tiffany C, Xu S, Dumont E, Janmohamed S. Design of Two Phase III, Randomized, Multicenter Studies Comparing Gepotidacin with Nitrofurantoin for the Treatment of Uncomplicated Urinary Tract Infection in Female Participants. Infect Dis Ther. 2022 Dec;11(6):2297-2310. doi: 10.1007/s40121-022-00706-9. Epub 2022 Oct 21. PMID 36271314
- [Derived] Fishman C, Caverly Rae JM, Posobiec LM, Laffan SB, Lerman SA, Pearson N, Janmohamed S, Dumont E, Nunn-Floyd D, Stanislaus DJ. Novel Bacterial Topoisomerase Inhibitor Gepotidacin Demonstrates Absence of Fluoroquinolone-Like Arthropathy in Juvenile Rats. Antimicrob Agents Chemother. 2022 Nov 15;66(11):e0048322. doi: 10.1128/aac.00483-22. Epub 2022 Oct 18. PMID 36255258
- [Derived] Scangarella-Oman NE, Hossain M, Hoover JL, Perry CR, Tiffany C, Barth A, Dumont EF. Dose Selection for Phase III Clinical Evaluation of Gepotidacin (GSK2140944) in the Treatment of Uncomplicated Urinary Tract Infections. Antimicrob Agents Chemother. 2022 Mar 15;66(3):e0149221. doi: 10.1128/AAC.01492-21. Epub 2022 Jan 3. PMID 34978887

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1605 unique participants were enrolled in the study including one participant that was randomized twice in error. This participant signed two different informed consent forms, therefore that participant was counted as enrolling twice.
Groups:
- Gepotidacin: Participants with uncomplicated urinary tract infection (uUTI) (acute cystitis) randomized to receive gepotidacin 1500 milligram (mg) (2*750 mg, tablets), twice daily (BID), orally on Day 1 to Day 5. The total daily dose of gepotidacin received was 3000 mg. Participants also received 1 capsule of placebo matched with nitrofurantoin BID, orally on Day 1 to Day 5. All doses were administered after food consumption and with water.
- Nitrofurantoin: Participants with uncomplicated urinary tract infection (acute cystitis) randomized to receive nitrofurantoin 100 mg capsule, BID, orally on Day 1 to Day 5. The total daily dose of nitrofurantoin received was 200 mg. Participants also received 2 tablets of placebo matched with gepotidacin BID, orally on Day 1 to Day 5. All doses were administered after food consumption and with water.
Period: Overall Study
Arm/Group | Gepotidacin | Nitrofurantoin
Started (Participants randomly assigned to the study treatment were included in Intent-to-Treat (ITT) population) | 805 | 800
Safety Population (Safety population included all randomized participants who receive at least 1 dose of study treatment.) | 804 | 798
Microbiological ITT (Micro ITT) Population (Microbiological ITT (micro-ITT) population included all participants randomly assigned to study treatment who receive at least 1 dose of study treatment and have a qualifying baseline uropathogen [10^5 CFU/mL] from a quantitative bacteriological culture of a pretreatment clean catch midstream urine specimen.) | 331 | 324
Micro-ITT NTF-S Population (Micro-ITT NTF-S population is defined as all participants in the micro-ITT population whose baseline qualifying uropathogens [10^5 CFU/mL] are all susceptible to nitrofurantoin (NTF-S).) | 292 | 275
Micro-ITT NTF-S (IA Set) Population (Microbiological intent-to-treat susceptible to nitrofurantoin (micro-ITT NTF-S) (IA Set) population included participants in the micro ITT NTF-S who per the interim analysis data had the opportunity to reach their Test of Cure (TOC) visit, or had not yet reached their TOC visit, but were already known to be failures.) | 277 | 264
Completed | 748 | 759
Not Completed | 57 | 41
Not completed — Lost to Follow-up | 12 | 11
Not completed — Withdrawal by Subject | 20 | 18
Not completed — Adverse Event | 19 | 4
Not completed — Physician Decision | 5 | 3
Not completed — Screening Failure due to creatinine clearance and body mass index | 0 | 1
Not completed — Protocol Deviation | 1 | 4

BASELINE CHARACTERISTICS:
Population: Participants randomly assigned to the study treatment were included in the ITT population.
Groups:
- Gepotidacin: Participants with uncomplicated urinary tract infection (acute cystitis) randomized to receive gepotidacin 1500 milligram (mg) (2*750 mg, tablets), twice daily (BID), orally on Day 1 to Day 5. The total daily dose of gepotidacin received was 3000 mg. Participants also received 1 capsule of placebo matched with nitrofurantoin BID, orally on Day 1 to Day 5. All doses were administered after food consumption and with water.
- Total: Total of all reporting groups
Arm/Group | Gepotidacin | Nitrofurantoin | Total
Number analyzed (Participants) | 805 | 800 | 1605
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.2 (17.84) | 48.4 (17.72) | 48.3 (17.77)
Age, Customized [Count of Participants; unit: Participants]
  Less than (<) 18 years | 8 | 3 | 11
  More than or equal to (>=) 18 years to 50 years | 427 | 430 | 857
  More than (>) 50 years | 370 | 367 | 737
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 805 | 800 | 1605
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 246 | 232 | 478
  Not Hispanic or Latino | 559 | 568 | 1127
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 51 | 65 | 116
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 74 | 62 | 136
  White | 674 | 668 | 1342
  More than one race | 2 | 4 | 6
  Unknown or Not Reported | 1 | 0 | 1
Baseline Acute Cystitis Recurrence [Count of Participants; unit: Participants] — Recurrent infection was defined as a confirmed infection with at least 1 episode within the past 3 months, at least 2 episodes within the past 6 months, or at least 3 episodes within the past 12 months before study entry.
  Participants
    Recurrent Infection | 334 | 338 | 672
    Non-Recurrent Infection | 471 | 462 | 933

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Therapeutic Response (TR) (Combined Per Participant Clinical and Microbiological Response) at the Test-of-Cure (TOC) Visit - Micro-ITT NTF-S (IA Set)
Description: TR at TOC (success/failure) is a measure of the overall efficacy response. A therapeutic success at TOC referred to participant who have been deemed both a microbiological success (reduction of all qualifying bacterial uropathogens recovered at Baseline [BL] to <10^3 colony forming units per milliliter [CFU/mL] without receiving other systemic antimicrobials [AB] before the TOC visit) and a clinical success (resolution of symptoms of acute cystitis present at BL and no symptoms without receiving other AB before the TOC visit [or AB for uUTI on day of TOC visit]). Lack of clinical or microbiological success (including missing outcome assessments) was considered as therapeutic failure.
Time Frame: TOC visit (Days 9 to 16)
Population: Microbiological intent-to-treat susceptible to nitrofurantoin - (Micro-ITT NTF-S) (Interim Analysis [IA] Set) population included participants in the micro ITT NTF-S who per the interim analysis data had the opportunity to reach their Test of Cure (TOC) visit, or had not yet reached their TOC visit, but were already known to be failures.
Measure: Count of Participants; unit: Participants
Arm/Group | Gepotidacin | Nitrofurantoin
Number analyzed (Participants) | 277 | 264
Participants
  Therapeutic Success | 162 | 115
  Therapeutic Failure | 115 | 149
Statistical Analysis 1: Comparison: Gepotidacin vs Nitrofurantoin; Test type: Non-Inferiority — The difference in success rate between treatment groups (gepotidacin - nitrofurantoin) was calculated using Miettinen-Nurminen Summary Score Method adjusted for age group and acute cystitis recurrence strata combinations. Criteria for non-inferiority is if the Z-statistic for non-inferiority is greater than the 2.098 Z-statistic boundary; Adjusted Difference in Percent = 14.6, 95% CI 2-sided [6.4 to 22.8]; Observed Z statistic value for Noninferiority was 5.8838
Statistical Analysis 2: Comparison: Gepotidacin vs Nitrofurantoin; The difference in success rate between treatment groups (gepotidacin - nitrofurantoin) was calculated using Miettinen-Nurminen Summary Score Method adjusted for age group and acute cystitis recurrence strata combinations. Criteria for superiority is if the one-sided p-value is less than the 0.018 p-value boundary; Test type: Superiority; p = 0.0003, 1-sided p-value for Test of Superiority; Adjusted difference in Percent = 14.6, 95% CI 2-sided [6.4 to 22.8]

2. Primary Outcome: Number of Participants With Therapeutic Response (TR) (Combined Per Participant Clinical and Microbiological Response) at the Test-of-Cure (TOC) Visit - Micro-ITT NTF-S Population
Description: TR at TOC (success/failure) is a measure of the overall efficacy response. A therapeutic success at TOC referred to participant who have been deemed both a microbiological success (reduction of all qualifying bacterial uropathogens recovered at Baseline [BL] to <10^3 colony forming units per milliliter [CFU/mL] without receiving other systemic antimicrobials [AB] before the TOC visit) and a clinical success (resolution of symptoms of acute cystitis present at BL and no new symptoms without receiving other AB before the TOC visit [or AB for uUTI on day of TOC visit]). Lack of clinical or microbiological success (including missing outcome assessments) was considered as therapeutic failure.
Time Frame: TOC visit (Days 9 to 16)
Population: Micro-ITT NTF-S population
Measure: Count of Participants; unit: Participants
Arm/Group | Gepotidacin | Nitrofurantoin
Number analyzed (Participants) | 292 | 275
Participants
  Therapeutic Success | 172 | 121
  Therapeutic Failure | 120 | 154

3. Secondary Outcome: Number of Participants With Clinical Outcome at the TOC Visit - Micro-ITT NTF-S Population
Description: Clinical outcomes at TOC were categorized as clinical resolution, clinical improvement, clinical worsening and unable to determine. Clinical resolution at TOC was defined as resolution of signs and symptoms of acute cystitis present at baseline (BL) (and no symptoms) without receiving any other AB before the TOC visit. Clinical improvement at TOC was defined as improvement (but not complete resolution) in total symptom score (CSS) from BL, without receiving any other AB before the TOC visit. Clinical worsening at TOC was defined as worsening or no change in CSS from BL or received other AB for the current infection (uUTI) before or on the date of the TOC visit. Unable to determine outcome criteria were: BL score is missing (and thus improvement/worsening cannot be determined), TOC assessment is missing, or receipt of other AB not for the current infection before the TOC visit (unless clinical worsening outcome criteria were met).
Time Frame: TOC visit (Days 9 to 16)
Population: Micro-ITT NTF-S population
Measure: Count of Participants; unit: Participants
Arm/Group | Gepotidacin | Nitrofurantoin
Number analyzed (Participants) | 292 | 275
Participants
  Clinical Resolution | 199 | 175
  Clinical Improvement (CI) | 51 | 68
  Clinical Worsening (CW) | 20 | 17
  Unable to Determine | 22 | 15

4. Secondary Outcome: Number of Participants With Clinical Response at the TOC Visit - Micro-ITT NTF-S Population
Description: Clinical response at TOC was categorized as clinical success and clinical failure. Clinical success at TOC was defined as resolution of symptoms of acute cystitis present at BL (and no new symptoms), without receiving any other AB before the TOC visit. Lack of resolution, including receipt of an AB for uUTI at the TOC visit, or a missing outcome assessment was defined as Clinical Failure at TOC.
Time Frame: TOC visit (Days 9 to 16)
Population: Micro-ITT NTF-S population.
Measure: Count of Participants; unit: Participants
Arm/Group | Gepotidacin | Nitrofurantoin
Number analyzed (Participants) | 292 | 275
Participants
  Clinical Success | 199 | 175
  Clinical Failure | 93 | 100

5. Secondary Outcome: Number of Participants With Microbiological Outcome (MO) at the TOC Visit - Micro-ITT NTF-S Population
Description: Participant-level MOs at TOC were categorized as microbiological eradication (ME), microbiological persistence (MP), microbiological recurrence (MR) and unable to determine (UTD). ME at TOC was defined as all baseline qualifying uropathogens (QUP) have an outcome of eradication at TOC (i.e., <10^3 CFU/mL without the participant receiving other systemic antimicrobials before the TOC Visit). MP at TOC was defined as at least 1 QUP has an outcome of persistence (≥10^3 CFU/mL) at TOC. MR at TOC was defined as at least 1 QUP had an outcome of recurrence and none have an outcome of persistence at TOC. UTD at TOC was defined as all QUP outcomes are UTD at TOC.
Time Frame: TOC Visit (Days 9 to 16)
Population: Micro-ITT NTF-S population.
Measure: Count of Participants; unit: Participants
Arm/Group | Gepotidacin | Nitrofurantoin
Number analyzed (Participants) | 292 | 275
Participants
  Microbiological Eradication (ME) | 213 | 158
  Microbiological Persistence (MP) | 13 | 31
  Microbiological Recurrence (MR) | 19 | 52
  Unable to Determine (UTD) | 47 | 34

6. Secondary Outcome: Number of Participants With Microbiological Response at the TOC Visit - Micro-ITT NTF-S Population
Description: Participant-level microbiological response at TOC was categorized as microbiological success and microbiological failure. Microbiological success at TOC was defined as all baseline qualifying uropathogens (QUP)s had a microbiological outcome of eradication at TOC visit. Microbiological failure was defined as lack of microbiological success, including those participants with UTD outcomes.
Time Frame: TOC visit (Days 9 to 16)
Population: Micro-ITT NTF-S population.
Measure: Count of Participants; unit: Participants
Arm/Group | Gepotidacin | Nitrofurantoin
Number analyzed (Participants) | 292 | 275
Participants
  Microbiological Success | 213 | 158
  Microbiological Failure | 79 | 117

7. Secondary Outcome: Number of Participants With Therapeutic Response (TR) (Combined Per Participant Clinical and Microbiological Response) at the Follow up (FU) Visit - Micro-ITT NTF-S Population
Description: TR at FU was categorized as therapeutic success and therapeutic failure. A therapeutic success at FU referred to participants who have been deemed both a microbiological success (reduction of all QUPs recovered at BL to <10^3 CFU/mL, following microbiological eradication at the TOC visit, without receiving other AB before the FU visit) and a clinical success (resolution of signs and symptoms of acute cystitis demonstrated at the TOC visit persist at the FU visit and no new signs and symptoms, without receiving other AB before the FU visit [or AB for uUTI on day of FU visit]). Lack of clinical or microbiological success (including missing outcome assessments) was considered as therapeutic failure.
Time Frame: FU visit (Days 21 to 31)
Population: Micro-ITT NTF-S population.
Measure: Count of Participants; unit: Participants
Arm/Group | Gepotidacin | Nitrofurantoin
Number analyzed (Participants) | 292 | 275
Participants
  Therapeutic Success | 126 | 95
  Therapeutic Failure | 166 | 180

8. Secondary Outcome: Number of Participants With Clinical Outcome at the Follow up (FU) Visit - Micro-ITT NTF-S Population
Description: Clinical outcomes at FU were categorized as SCR, DCR, CI, CW, CR and UTD. SCR at FU was resolution of symptoms of acute cystitis demonstrated at the TOC persist at the FU (and no symptoms), without receiving other AB before the FU. DCR at FU was resolution of symptoms of acute cystitis present at BL after clinical failure at TOC without receiving AB before FU. CI at FU was improvement in CSS from BL, but not complete resolution without receiving AB before FU. CW at FU was worsening or no change in CSS at FU compared to BL after clinical failure at TOC or receiving other AB for the current infection (uUTI) before or on the date of the FU. CR at FU was symptoms of acute cystitis reoccur at FU after clinical success at TOC. Unable to determine outcome criteria at FU were BL score missing, FU assessment missing or received other AB not for the current infection (uUTI) prior to the assessment (unless CS or CR outcome criteria were met).
Time Frame: FU visit (Days 21 to 31)
Population: Micro-ITT NTF-S population
Measure: Count of Participants; unit: Participants
Arm/Group | Gepotidacin | Nitrofurantoin
Number analyzed (Participants) | 292 | 275
Participants
  Sustained Clinical Resolution (SCR) | 168 | 154
  Delayed Clinical Resolution (DCR) | 34 | 35
  Clinical Improvement (CI) | 15 | 19
  Clinical Worsening (CW) | 26 | 32
  Clinical Recurrence (CR) | 8 | 7
  Unable to Determine (UTD) | 41 | 28

9. Secondary Outcome: Number of Participants With Clinical Response at the Follow up (FU) Visit - Micro-ITT NTF-S Population
Description: Clinical response at FU was categorized as clinical success and clinical failure. Clinical success at FU was defined as resolution of symptoms of acute cystitis demonstrated at TOC persist at the FU visit (and no new symptoms), without receiving other AB before the FU visit. Lack of sustained clinical resolution or a missing outcome assessment was defined as clinical failure.
Time Frame: FU visit (Days 21 to 31)
Population: Micro-ITT NTF-S population
Measure: Count of Participants; unit: Participants
Arm/Group | Gepotidacin | Nitrofurantoin
Number analyzed (Participants) | 292 | 275
Participants
  Clinical Success | 168 | 154
  Clinical Failure | 124 | 121

10. Secondary Outcome: Number of Participants With Microbiological Outcome (MO) at the Follow up (FU) Visit - Micro-ITT NTF-S Population
Description: Participant-level MOs at FU were categorized as sustained microbiological eradication (SME), microbiological recurrence (MR), microbiological persistence (MP), delayed microbiological eradication (DME) and unable to determine (UTD). SME at FU was defined as all baseline QUPs had an outcome of sustained eradication at FU (i.e., <10^3 CFU/mL without the participant receiving other systemic antimicrobials before the FU Visit). MR at FU was defined as at least one QUP had an outcome of recurrence (≥10^3 CFU/mL) and none had an outcome of persistence at FU. MP at FU was defined as at least one QUP had an outcome of persistence at FU. DME at FU was defined as at least one QUP had an outcome of delayed eradication and none had an outcome of persistence or recurrence at FU. UTD at FU was defined as all QUP outcomes were unable to determine at FU.
Time Frame: FU visit (Days 21 to 31)
Population: Micro-ITT NTF-S population.
Measure: Count of Participants; unit: Participants
Arm/Group | Gepotidacin | Nitrofurantoin
Number analyzed (Participants) | 292 | 275
Participants
  Sustained Microbiological Eradication (SME) | 154 | 119
  Microbiological Persistence (MP) | 19 | 44
  Microbiological Recurrence (MR) | 29 | 23
  Delayed Microbiological Eradication (DME) | 20 | 28
  Unable to Determine (UTD) | 70 | 61

11. Secondary Outcome: Number of Participants With Microbiological Response at the Follow up (FU) Visit - Micro-ITT NTF-S Population
Description: Participant- level microbiological response at FU was categorized as microbiological success and microbiological failure. Microbiological success at FU was defined as all baseline QUPs had a microbiological outcome of sustained eradication at FU visit. Microbiological failure at FU was defined as not meeting criteria of microbiological success including those participants with UTD outcome.
Time Frame: FU visit (Days 21 to 31)
Population: Micro-ITT NTF-S population.
Measure: Count of Participants; unit: Participants
Arm/Group | Gepotidacin | Nitrofurantoin
Number analyzed (Participants) | 292 | 275
Participants
  Microbiological Success | 154 | 119
  Microbiological Failure | 138 | 156

12. Secondary Outcome: Number of Participants With Clinical Outcome at the TOC Visit - Intent-to-Treat (ITT) Population
Description: Clinical outcomes at TOC were categorized as clinical resolution, clinical improvement, clinical worsening and unable to determine. Clinical resolution at TOC was defined as resolution symptoms of acute cystitis present at baseline (BL) (and no symptoms) without receiving any other AB before the TOC visit. Clinical improvement at TOC was defined as improvement (but not complete resolution) in CSS from BL, without receiving any other AB before the TOC visit. Clinical worsening at TOC was defined as worsening or no change in CSS from BL or received other AB for the current infection (uUTI) before or on the date of the TOC visit. Unable to determine outcome criteria were: BL score is missing (and thus improvement/worsening cannot be determined), TOC assessment is missing, or receipt of other AB not for the current infection before the TOC visit (unless clinical worsening outcome criteria were met).
Time Frame: TOC visit (Days 9 to 16)
Population: Intent-to-Treat (ITT) population included all participants randomly assigned to study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Gepotidacin | Nitrofurantoin
Number analyzed (Participants) | 805 | 800
Participants
  Clinical Resolution | 549 | 517
  Clinical Improvement | 153 | 199
  Clinical Worsening | 36 | 39
  Unable to Determine | 67 | 45

13. Secondary Outcome: Number of Participants With Clinical Response at the TOC Visit - Intent-to-Treat (ITT) Population
Description: Clinical response at TOC was categorized as clinical success and clinical failure. Clinical success at TOC was defined as resolution of signs and symptoms of acute cystitis present at BL (and no new symptoms), without receiving any other AB before the TOC visit. Lack of resolution, including receipt of an AB for uUTI at the TOC visit, or a missing outcome assessment was defined as Clinical Failure.
Time Frame: TOC visit (Days 9 to 16)
Population: Intent-to-Treat (ITT) population
Measure: Count of Participants; unit: Participants
Arm/Group | Gepotidacin | Nitrofurantoin
Number analyzed (Participants) | 805 | 800
Participants
  Clinical Success | 549 | 517
  Clinical Failure | 256 | 283

14. Secondary Outcome: Number of Participants With Clinical Outcome at the Follow up (FU) Visit - Intent-to-Treat (ITT) Population
Description: Clinical outcomes at FU were categorized as Sustained Clinical Response (SCR), Delayed Clinical Response (DCR), CI, CW, Clinical Recurrence (CR) and UTD. SCR at FU was resolution of symptoms of acute cystitis demonstrated at TOC persist at the FU (and no symptoms), without receiving other AB before the FU. DCR at FU was resolution of symptoms of acute cystitis present at BL after clinical failure at TOC without receiving AB before FU. CI at FU was improvement in CSS from BL, but not complete resolution without receiving AB before FU. CW at FU was worsening or no change in CSS at FU compared to BL after clinical failure at TOC or receiving other AB for the current infection (uUTI) before or on the date of the FU. CR at FU was symptoms of acute cystitis reoccur at FU after clinical success at TOC. UTD outcome criteria at FU were BL score missing, FU assessment missing or received other AB not for current infection (uUTI) prior to assessment (unless CS or CR outcome criteria were met).
Time Frame: FU visit (Days 21 to 31)
Population: Intent-to-Treat (ITT) population
Measure: Count of Participants; unit: Participants
Arm/Group | Gepotidacin | Nitrofurantoin
Number analyzed (Participants) | 805 | 800
Participants
  Sustained Clinical Resolution (SCR) | 478 | 443
  Delayed Clinical Resolution (DCR) | 108 | 116
  Clinical Improvement (CI) | 40 | 52
  Clinical Worsening (CW) | 51 | 65
  Clinical Recurrence (CR) | 25 | 28
  Unable to Determine (UTD) | 103 | 96

15. Secondary Outcome: Number of Participants With Clinical Response at the Follow up (FU) Visit - Intent-to-Treat (ITT) Population
Description: as for outcome 9
Time Frame: FU visit (Days 21 to 31)
Population: Intent-to-Treat (ITT) population
Measure: Count of Participants; unit: Participants
Arm/Group | Gepotidacin | Nitrofurantoin
Number analyzed (Participants) | 805 | 800
Participants
  Clinical Success | 478 | 443
  Clinical Failure | 327 | 357

16. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study treatment.
Time Frame: From the time of first dose (Day 1) through the final follow-up visit (Day 21-31)
Population: Safety population included all randomized participants who receive at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Gepotidacin | Nitrofurantoin
Number analyzed (Participants) | 804 | 798
Participants | 285 | 200

17. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: An SAE is defined as any untoward medical occurrence that, at any dose may result in death or is life-threatening or requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity or is a congenital anomaly/birth defect or any other situation according to medical or scientific judgment or is associated with liver injury and impaired liver function.
Time Frame: From the time of first dose (Day 1) through the final follow-up visit (Day 21-31)
Population: Safety population included all randomized participants who receive at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Gepotidacin | Nitrofurantoin
Number analyzed (Participants) | 804 | 798
Participants | 5 | 5

18. Secondary Outcome: Change From Baseline in Hematology Parameters: Neutrophil Count, Lymphocyte Count, Monocyte Count, Eosinophil Count, Basophil Count and Platelet Count at On Therapy and Test of Cure Visit
Description: Blood samples were collected for the analysis of hematology parameters: neutrophil count, lymphocyte count, monocyte count, eosinophil count, basophil count and platelet count. Baseline is defined as the latest pre-dose assessment with a non-missing value.
Time Frame: Baseline (on or before Day 1), On-Therapy (Days 2 to 5), and Test of cure (Days 9 to 16)
Population: Safety population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Giga cells per Liter (10^9 cells/L)
Arm/Group | Gepotidacin | Nitrofurantoin
Number analyzed (Participants) | 736 | 737
Giga cells per Liter (10^9 cells/L)
  Eosinophils, Baseline: number analyzed (Participants) | 702 | 698
  Eosinophils, Baseline | 0.161 (0.1350) | 0.163 (0.1331)
  Eosinophils, On-Therapy: number analyzed (Participants) | 622 | 606
  Eosinophils, On-Therapy | 0.006 (0.0841) | 0.013 (0.0814)
  Eosinophils, Test of Cure: number analyzed (Participants) | 608 | 599
  Eosinophils, Test of Cure | 0.015 (0.0906) | 0.018 (0.1081)
  Basophils, Baseline: number analyzed (Participants) | 642 | 668
  Basophils, Baseline | 0.054 (0.0227) | 0.053 (0.0228)
  Basophils, On-Therapy: number analyzed (Participants) | 533 | 550
  Basophils, On-Therapy | -0.001 (0.0195) | 0.001 (0.0194)
  Basophils, Test of Cure: number analyzed (Participants) | 528 | 551
  Basophils, Test of Cure | 0.000 (0.0209) | 0.001 (0.0183)
  Lymphocytes, Baseline | 2.091 (0.6954) | 2.121 (0.7122)
  Lymphocytes, On-Therapy: number analyzed (Participants) | 661 | 657
  Lymphocytes, On-Therapy | -0.018 (0.4523) | -0.076 (0.5051)
  Lymphocytes, Test of Cure: number analyzed (Participants) | 641 | 651
  Lymphocytes, Test of Cure | -0.010 (0.5292) | 0.059 (0.5839)
  Monocytes, Baseline | 0.529 (0.1803) | 0.525 (0.1790)
  Monocytes, On-Therapy: number analyzed (Participants) | 661 | 657
  Monocytes, On-Therapy | -0.020 (0.1487) | 0.003 (0.1711)
  Monocytes, Test of Cure: number analyzed (Participants) | 641 | 651
  Monocytes, Test of Cure | -0.029 (0.1731) | -0.012 (0.1778)
  Neutrophils, Baseline | 4.582 (1.8893) | 4.755 (1.8821)
  Neutrophils, On-Therapy: number analyzed (Participants) | 661 | 656
  Neutrophils, On-Therapy | -0.490 (1.6201) | -0.453 (1.7453)
  Neutrophils, Test of Cure: number analyzed (Participants) | 641 | 651
  Neutrophils, Test of Cure | -0.534 (2.0207) | -0.494 (1.9072)
  Platelets, Baseline: number analyzed (Participants) | 723 | 729
  Platelets, Baseline | 280.3 (68.46) | 287.2 (73.51)
  Platelets, On-Therapy: number analyzed (Participants) | 649 | 648
  Platelets, On-Therapy | -1.1 (33.03) | -2.5 (36.67)
  Platelets, Test of Cure: number analyzed (Participants) | 626 | 637
  Platelets, Test of Cure | 6.8 (42.12) | 5.5 (58.04)

19. Secondary Outcome: Change From Baseline in Hematology Parameter: Hemoglobin Level
Description: Blood samples were collected for the analysis of hemoglobin level. Baseline is defined as the latest pre-dose assessment with a non-missing value.
Time Frame: Baseline (on or before Day 1), On-Therapy (Days 2 to 5), and Test of cure (Days 9 to 16)
Population: Safety population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Gram per Liter (g/L)
Arm/Group | Gepotidacin | Nitrofurantoin
Number analyzed (Participants) | 739 | 737
Gram per Liter (g/L)
  Baseline | 132.5 (13.25) | 131.7 (14.28)
  On-Therapy: number analyzed (Participants) | 665 | 657
  On-Therapy | -1.5 (6.74) | -1.9 (6.82)
  Test of Cure: number analyzed (Participants) | 643 | 653
  Test of Cure | -1.3 (7.44) | -1.4 (8.33)

20. Secondary Outcome: Change From Baseline in Hematology Parameter: Hematocrit Level
Description: Blood samples were collected for the analysis of hematocrit level. Baseline is defined as the latest pre-dose assessment with a non-missing value.
Time Frame: Baseline (on or before Day 1), On-Therapy (Days 2 to 5), and Test of cure (Days 9 to 16)
Population: Safety population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Percentage of hematocrit
Arm/Group | Gepotidacin | Nitrofurantoin
Number analyzed (Participants) | 739 | 737
Percentage of hematocrit
  Baseline | 0.4314 (0.04146) | 0.4292 (0.04348)
  On-Therapy: number analyzed (Participants) | 665 | 657
  On-Therapy | -0.0033 (0.02832) | -0.0041 (0.02715)
  Test of Cure: number analyzed (Participants) | 643 | 653
  Test of Cure | -0.0045 (0.02806) | -0.0029 (0.03194)

21. Secondary Outcome: Change From Baseline in Hematology Parameter: Erythrocytes (RBC) Count
Description: Blood samples were collected for the analysis of erythrocytes count. Baseline is defined as the latest pre-dose assessment with a non-missing value.
Time Frame: Baseline (on or before Day 1), On-Therapy (Days 2 to 5), and Test of cure (Days 9 to 16)
Population: Safety population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Tera cells per Liter (10^12 cells/L)
Arm/Group | Gepotidacin | Nitrofurantoin
Number analyzed (Participants) | 739 | 737
Tera cells per Liter (10^12 cells/L)
  Baseline | 4.539 (0.4211) | 4.539 (0.4379)
  On-Therapy: number analyzed (Participants) | 665 | 657
  On-Therapy | -0.046 (0.2309) | -0.060 (0.2513)
  Test of Cure: number analyzed (Participants) | 643 | 653
  Test of Cure | -0.038 (0.2634) | -0.049 (0.3052)

22. Secondary Outcome: Change From Baseline in Hematology Parameter: Mean Corpuscular Hemoglobin (MCH)
Description: Blood samples were collected for the analysis of MCH. Baseline is defined as the latest pre-dose assessment with a non-missing value.
Time Frame: Baseline (on or before Day 1), On-Therapy (Days 2 to 5), and Test of cure (Days 9 to 16)
Population: Safety population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Picogram (pg)
Arm/Group | Gepotidacin | Nitrofurantoin
Number analyzed (Participants) | 739 | 737
Picogram (pg)
  Baseline | 29.28 (2.537) | 29.09 (2.644)
  On-Therapy: number analyzed (Participants) | 665 | 657
  On-Therapy | -0.02 (0.795) | -0.02 (0.820)
  Test of Cure: number analyzed (Participants) | 643 | 653
  Test of Cure | -0.04 (0.780) | 0.02 (0.917)

23. Secondary Outcome: Change From Baseline in Hematology Parameter: Mean Corpuscular Volume (MCV)
Description: Blood samples were collected for the analysis of MCV. Baseline is defined as the latest pre-dose assessment with a non-missing value.
Time Frame: Baseline (on or before Day 1), On-Therapy (Days 2 to 5), and Test of cure (Days 9 to 16)
Population: Safety population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Femtolitre (fL)
Arm/Group | Gepotidacin | Nitrofurantoin
Number analyzed (Participants) | 739 | 737
Femtolitre (fL)
  Baseline | 95.30 (7.191) | 94.82 (7.511)
  On-Therapy: number analyzed (Participants) | 665 | 657
  On-Therapy | 0.26 (4.287) | 0.35 (4.303)
  Test of Cure: number analyzed (Participants) | 643 | 653
  Test of Cure | -0.15 (4.049) | 0.39 (4.730)

24. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters: Serum Blood Urea Nitrogen (BUN), Glucose Non-fasting, Calcium, Chloride, Sodium, Magnesium, Phosphate, and Potassium Levels
Description: Blood samples were collected for the analysis of clinical chemistry parameters. Baseline is defined as the latest pre-dose assessment with a non-missing value.
Time Frame: Baseline (on or before Day 1), On-Therapy (Days 2 to 5), and Test of cure (Days 9 to 16)
Population: Safety population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: millimoles per liter (mmol/L)
Arm/Group | Gepotidacin | Nitrofurantoin
Number analyzed (Participants) | 781 | 777
millimoles per liter (mmol/L)
  Serum Urea Nitrogen, Baseline: number analyzed (Participants) | 780 | 776
  Serum Urea Nitrogen, Baseline | 4.742 (2.1107) | 4.724 (1.8645)
  Serum Urea Nitrogen, On- Therapy: number analyzed (Participants) | 714 | 721
  Serum Urea Nitrogen, On- Therapy | -0.056 (1.4269) | -0.018 (1.1663)
  Serum Urea Nitrogen, Test of Cure: number analyzed (Participants) | 703 | 716
  Serum Urea Nitrogen, Test of Cure | 0.022 (1.4000) | 0.131 (1.4826)
  Serum Calcium, Baseline: number analyzed (Participants) | 776 | 773
  Serum Calcium, Baseline | 2.363 (0.1196) | 2.362 (0.1083)
  Serum Calcium, On-Therapy: number analyzed (Participants) | 705 | 717
  Serum Calcium, On-Therapy | -0.010 (0.0950) | -0.018 (0.0944)
  Serum Calcium, Test of Cure: number analyzed (Participants) | 698 | 712
  Serum Calcium, Test of Cure | -0.014 (0.1070) | -0.016 (0.0981)
  Serum Chloride, Baseline: number analyzed (Participants) | 780 | 776
  Serum Chloride, Baseline | 101.0 (3.27) | 100.9 (3.27)
  Serum Chloride, On-Therapy: number analyzed (Participants) | 713 | 721
  Serum Chloride, On-Therapy | 0.3 (2.80) | 0.1 (2.85)
  Serum Chloride, Test of Cure: number analyzed (Participants) | 701 | 716
  Serum Chloride, Test of Cure | 0.4 (2.93) | 0.4 (3.02)
  Serum Glucose, Baseline: number analyzed (Participants) | 777 | 774
  Serum Glucose, Baseline | 5.590 (1.9980) | 5.719 (2.1915)
  Serum Glucose, On-Therapy: number analyzed (Participants) | 705 | 719
  Serum Glucose, On-Therapy | 0.230 (1.5120) | 0.328 (1.9380)
  Serum Glucose, Test of Cure: number analyzed (Participants) | 698 | 709
  Serum Glucose, Test of Cure | 0.215 (1.4412) | 0.266 (1.6667)
  Serum Magnesium, Baseline: number analyzed (Participants) | 776 | 773
  Serum Magnesium, Baseline | 0.839 (0.0749) | 0.835 (0.0802)
  Serum Magnesium, On-Therapy: number analyzed (Participants) | 706 | 717
  Serum Magnesium, On-Therapy | -0.001 (0.0635) | -0.015 (0.0616)
  Serum Magnesium, Test of Cure: number analyzed (Participants) | 698 | 712
  Serum Magnesium, Test of Cure | -0.011 (0.0674) | -0.015 (0.0689)
  Serum Potassium, Baseline: number analyzed (Participants) | 776 | 772
  Serum Potassium, Baseline | 4.32 (0.414) | 4.27 (0.415)
  Serum Potassium, On-Therapy: number analyzed (Participants) | 701 | 717
  Serum Potassium, On-Therapy | -0.04 (0.417) | -0.03 (0.428)
  Serum Potassium, Test of Cure: number analyzed (Participants) | 696 | 710
  Serum Potassium, Test of Cure | -0.03 (0.438) | 0.00 (0.461)
  Serum Phosphate, Baseline: number analyzed (Participants) | 778 | 774
  Serum Phosphate, Baseline | 1.141 (0.1828) | 1.139 (0.1725)
  Serum Phosphate, On-Therapy: number analyzed (Participants) | 704 | 719
  Serum Phosphate, On-Therapy | -0.005 (0.1782) | -0.027 (0.1836)
  Serum Phosphate, Test of Cure: number analyzed (Participants) | 699 | 711
  Serum Phosphate, Test of Cure | 0.002 (0.1851) | -0.004 (0.1939)
  Serum Sodium, Baseline | 138.8 (2.64) | 138.8 (2.76)
  Serum Sodium, On-Therapy: number analyzed (Participants) | 714 | 724
  Serum Sodium, On-Therapy | 0.0 (2.64) | -0.2 (2.64)
  Serum Sodium, Test of Cure: number analyzed (Participants) | 702 | 717
  Serum Sodium, Test of Cure | 0.2 (2.91) | 0.1 (2.91)

25. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters: Total Bilirubin, Direct Bilirubin and Creatinine Levels
Description: as for outcome 24
Time Frame: Baseline (on or before Day 1), On-Therapy (Days 2 to 5), and Test of cure (Days 9 to 16)
Population: Safety population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: micromoles per Liter (umol/L)
Arm/Group | Gepotidacin | Nitrofurantoin
Number analyzed (Participants) | 779 | 776
micromoles per Liter (umol/L)
  Serum Direct Bilirubin, Baseline: number analyzed (Participants) | 93 | 84
  Serum Direct Bilirubin, Baseline | 4.61 (1.669) | 4.47 (1.128)
  Serum Direct Bilirubin, On- Therapy: number analyzed (Participants) | 50 | 41
  Serum Direct Bilirubin, On- Therapy | -0.18 (1.192) | -0.18 (1.114)
  Serum Direct Bilirubin, Test of Cure: number analyzed (Participants) | 46 | 38
  Serum Direct Bilirubin, Test of Cure | -0.19 (1.059) | 0.15 (1.288)
  Serum Total Bilirubin, Baseline: number analyzed (Participants) | 751 | 742
  Serum Total Bilirubin, Baseline | 6.57 (3.940) | 6.56 (3.518)
  Serum Total Bilirubin, On-Therapy: number analyzed (Participants) | 655 | 670
  Serum Total Bilirubin, On-Therapy | -0.28 (2.510) | -0.42 (2.672)
  Serum Total Bilirubin, Test of Cure: number analyzed (Participants) | 652 | 656
  Serum Total Bilirubin, Test of Cure | -0.01 (2.976) | -0.29 (3.230)
  Serum Creatinine, Baseline | 58.8 (30.59) | 58.1 (17.22)
  Serum Creatinine, On-Therapy: number analyzed (Participants) | 712 | 721
  Serum Creatinine, On-Therapy | 0.8 (30.31) | 0.3 (10.31)
  Serum Creatinine, Test of Cure: number analyzed (Participants) | 703 | 715
  Serum Creatinine, Test of Cure | 1.7 (14.00) | 1.5 (13.40)

26. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters: Albumin and Protein Levels
Description: as for outcome 24
Time Frame: Baseline (on or before Day 1), On-Therapy (Days 2 to 5), and Test of cure (Days 9 to 16)
Population: Safety population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: gram per Liter (g/L)
Arm/Group | Gepotidacin | Nitrofurantoin
Number analyzed (Participants) | 781 | 777
gram per Liter (g/L)
  Serum Albumin, Baseline | 45.2 (3.33) | 45.2 (3.11)
  Serum Albumin, On-Therapy: number analyzed (Participants) | 715 | 725
  Serum Albumin, On-Therapy | -0.4 (2.38) | -0.8 (2.56)
  Serum Albumin, Test of Cure: number analyzed (Participants) | 705 | 720
  Serum Albumin, Test of Cure | -0.5 (2.65) | -0.6 (2.84)
  Serum Protein, Baseline: number analyzed (Participants) | 778 | 774
  Serum Protein, Baseline | 71.5 (5.12) | 71.6 (4.72)
  Serum Protein, On-Therapy: number analyzed (Participants) | 709 | 719
  Serum Protein, On-Therapy | -0.7 (3.71) | -1.2 (3.89)
  Serum Protein, Test of Cure: number analyzed (Participants) | 700 | 711
  Serum Protein, Test of Cure | -1.0 (4.19) | -1.1 (4.32)

27. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters: Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT) and Alkaline Phosphatase (ALP) Levels
Description: as for outcome 24
Time Frame: Baseline (on or before Day 1), On-Therapy (Days 2 to 5), and Test of cure (Days 9 to 16)
Population: Safety population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Units per Liter (U/L)
Arm/Group | Gepotidacin | Nitrofurantoin
Number analyzed (Participants) | 777 | 774
Units per Liter (U/L)
  Serum ALT, Baseline: number analyzed (Participants) | 776 | 773
  Serum ALT, Baseline | 20.3 (20.34) | 19.5 (14.66)
  Serum ALT, On-Therapy: number analyzed (Participants) | 705 | 716
  Serum ALT, On-Therapy | 0.2 (10.8) | -0.1 (7.9)
  Serum ALT, Test of Cure: number analyzed (Participants) | 699 | 710
  Serum ALT, Test of Cure | 0.4 (15.81) | -0.2 (9.93)
  Serum AST, Baseline | 21.0 (13.72) | 20.2 (10.48)
  Serum AST, On-Therapy: number analyzed (Participants) | 706 | 719
  Serum AST, On-Therapy | 0.1 (9.83) | 0.0 (7.90)
  Serum AST, Test of Cure: number analyzed (Participants) | 700 | 710
  Serum AST, Test of Cure | 0.9 (9.89) | -0.5 (8.29)
  Serum ALP, Baseline: number analyzed (Participants) | 776 | 773
  Serum ALP, Baseline | 81.4 (29.96) | 81.7 (28.99)
  Serum ALP, On- Therapy: number analyzed (Participants) | 707 | 717
  Serum ALP, On- Therapy | -0.5 (9.61) | -0.1 (12.91)
  Serum ALP, Test of Cure: number analyzed (Participants) | 698 | 712
  Serum ALP, Test of Cure | -1.0 (12.00) | -0.4 (15.38)

28. Secondary Outcome: Number of Participants With Urinalysis Dipstick Results
Description: Urine samples were collected for urinalysis: Urine Glucose (GLU), Urine Protein (PRO), Urine Occult Blood (BLO), Urine Ketones (KET), Urine Nitrite (NIT) and Urine Leukocyte Esterase (LEU). Baseline is defined as the latest pre-dose assessment with a non-missing value. The dipstick test gives results in a semi-quantitative manner, and results can be read as Negative, Trace, Small, Moderate, Large, Positive, 50 milligram per deciliter (mg/dL), 150 mg/dL, >=500 mg/dL, 30 mg/dL, 100 mg/dL, 200 mg/dL, 5 mg/dL, 20 mg/dL, >=80 mg/dL indicating concentrations in the urine sample. In the row title (GLU, Baseline, Negative), GLU indicates parameter, Baseline is the visit and Negative indicates the concentration in the urine sample. Data is presented in similar way for others parameters.
Time Frame: Baseline (on or before Day 1), On-Therapy (Days 2 to 5), and Test of cure (Days 9 to 16)
Population: Safety population. Only those participants with data available at the specified data points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Gepotidacin | Nitrofurantoin
Number analyzed (Participants) | 789 | 783
Participants
  GLU, Baseline, Negative: number analyzed (Participants) | 779 | 773
  GLU, Baseline, Negative | 751 | 738
  GLU, Baseline, 50 mg/dL: number analyzed (Participants) | 779 | 773
  GLU, Baseline, 50 mg/dL | 4 | 5
  GLU, Baseline, 150 mg/dL: number analyzed (Participants) | 779 | 773
  GLU, Baseline, 150 mg/dL | 3 | 4
  GLU, Baseline, >= 500 mg/dL: number analyzed (Participants) | 779 | 773
  GLU, Baseline, >= 500 mg/dL | 21 | 26
  GLU, On-Therapy, Negative: number analyzed (Participants) | 731 | 737
  GLU, On-Therapy, Negative | 700 | 697
  GLU, On-Therapy, 50 mg/dL: number analyzed (Participants) | 731 | 737
  GLU, On-Therapy, 50 mg/dL | 7 | 7
  GLU, On-Therapy, 150 mg/dL: number analyzed (Participants) | 731 | 737
  GLU, On-Therapy, 150 mg/dL | 1 | 5
  GLU, On-Therapy, >= 500 mg/dL: number analyzed (Participants) | 731 | 737
  GLU, On-Therapy, >= 500 mg/dL | 23 | 28
  GLU, Test of Cure, Negative: number analyzed (Participants) | 719 | 727
  GLU, Test of Cure, Negative | 686 | 693
  GLU, Test of Cure, 50 mg/dL: number analyzed (Participants) | 719 | 727
  GLU, Test of Cure, 50 mg/dL | 9 | 10
  GLU, Test of Cure, 150 mg/dL: number analyzed (Participants) | 719 | 727
  GLU, Test of Cure, 150 mg/dL | 12 | 4
  GLU, Test of Cure, >= 500 mg/dL: number analyzed (Participants) | 719 | 727
  GLU, Test of Cure, >= 500 mg/dL | 12 | 20
  PRO, Baseline, Negative: number analyzed (Participants) | 778 | 769
  PRO, Baseline, Negative | 524 | 529
  PRO, Baseline, 30 mg/dL: number analyzed (Participants) | 778 | 769
  PRO, Baseline, 30 mg/dL | 171 | 149
  PRO, Baseline, 100 mg/dL: number analyzed (Participants) | 778 | 769
  PRO, Baseline, 100 mg/dL | 78 | 85
  PRO, Baseline, >=500 mg/dL: number analyzed (Participants) | 778 | 769
  PRO, Baseline, >=500 mg/dL | 5 | 6
  PRO, On-Therapy, Negative: number analyzed (Participants) | 731 | 737
  PRO, On-Therapy, Negative | 575 | 631
  PRO, On-Therapy, 30 mg/dL: number analyzed (Participants) | 731 | 737
  PRO, On-Therapy, 30 mg/dL | 110 | 83
  PRO, On-Therapy, 100 mg/dL: number analyzed (Participants) | 719 | 727
  PRO, On-Therapy, 100 mg/dL | 43 | 19
  PRO, On-Therapy, >=500 mg/dL: number analyzed (Participants) | 731 | 737
  PRO, On-Therapy, >=500 mg/dL | 3 | 4
  PRO, Test of Cure, Negative: number analyzed (Participants) | 719 | 727
  PRO, Test of Cure, Negative | 605 | 605
  PRO, Test of Cure, 30 mg/dL: number analyzed (Participants) | 719 | 727
  PRO, Test of Cure, 30 mg/dL | 88 | 88
  PRO, Test of Cure, 100 mg/dL: number analyzed (Participants) | 731 | 737
  PRO, Test of Cure, 100 mg/dL | 25 | 34
  PRO, Test of Cure, >=500 mg/dL: number analyzed (Participants) | 719 | 727
  PRO, Test of Cure, >=500 mg/dL | 1 | 0
  BLO, Baseline, Positive: number analyzed (Participants) | 784 | 777
  BLO, Baseline, Positive | 0 | 2
  BLO, Baseline, Negative: number analyzed (Participants) | 784 | 777
  BLO, Baseline, Negative | 345 | 348
  BLO, Baseline, Trace: number analyzed (Participants) | 784 | 777
  BLO, Baseline, Trace | 2 | 0
  BLO, Baseline, Small: number analyzed (Participants) | 784 | 777
  BLO, Baseline, Small | 229 | 217
  BLO, Baseline, Moderate: number analyzed (Participants) | 784 | 777
  BLO, Baseline, Moderate | 128 | 129
  BLO, Baseline, Large: number analyzed (Participants) | 784 | 777
  BLO, Baseline, Large | 80 | 81
  BLO, On-Therapy, Negative: number analyzed (Participants) | 731 | 737
  BLO, On-Therapy, Negative | 560 | 520
  BLO, On-Therapy, Small: number analyzed (Participants) | 731 | 737
  BLO, On-Therapy, Small | 116 | 161
  BLO, On-Therapy, Moderate: number analyzed (Participants) | 731 | 737
  BLO, On-Therapy, Moderate | 23 | 30
  BLO, On-Therapy, Large: number analyzed (Participants) | 731 | 737
  BLO, On-Therapy, Large | 32 | 26
  BLO, Test of Cure, Negative: number analyzed (Participants) | 719 | 727
  BLO, Test of Cure, Negative | 517 | 511
  BLO, Test of Cure, Small: number analyzed (Participants) | 719 | 727
  BLO, Test of Cure, Small | 128 | 139
  BLO, Test of Cure, Moderate: number analyzed (Participants) | 719 | 727
  BLO, Test of Cure, Moderate | 49 | 45
  BLO, Test of Cure, Large: number analyzed (Participants) | 719 | 727
  BLO, Test of Cure, Large | 25 | 32
  KET, Baseline, Negative: number analyzed (Participants) | 779 | 773
  KET, Baseline, Negative | 754 | 748
  KET, Baseline, 5 mg/dL: number analyzed (Participants) | 779 | 773
  KET, Baseline, 5 mg/dL | 14 | 18
  KET, Baseline, 20 mg/dL: number analyzed (Participants) | 779 | 773
  KET, Baseline, 20 mg/dL | 11 | 7
  KET, On-Therapy, Negative: number analyzed (Participants) | 731 | 737
  KET, On-Therapy, Negative | 712 | 699
  KET, On-Therapy, 5 mg/dL: number analyzed (Participants) | 731 | 737
  KET, On-Therapy, 5 mg/dL | 14 | 22
  KET, On-Therapy, 20 mg/dL: number analyzed (Participants) | 731 | 737
  KET, On-Therapy, 20 mg/dL | 5 | 15
  KET, On-Therapy, >=80 mg/dL: number analyzed (Participants) | 731 | 737
  KET, On-Therapy, >=80 mg/dL | 0 | 1
  KET, Test of Cure, Negative: number analyzed (Participants) | 719 | 727
  KET, Test of Cure, Negative | 706 | 700
  KET, Test of Cure, 5 mg/dL: number analyzed (Participants) | 719 | 727
  KET, Test of Cure, 5 mg/dL | 7 | 20
  KET, Test of Cure, 20 mg/dL: number analyzed (Participants) | 719 | 727
  KET, Test of Cure, 20 mg/dL | 6 | 7
  NIT, Baseline, Negative | 552 | 531
  NIT, Baseline, Positive | 237 | 252
  NIT, On-Therapy, Negative: number analyzed (Participants) | 731 | 737
  NIT, On-Therapy, Negative | 694 | 697
  NIT, On-Therapy, Positive: number analyzed (Participants) | 731 | 737
  NIT, On-Therapy, Positive | 37 | 40
  NIT, Test of Cure, Negative: number analyzed (Participants) | 719 | 727
  NIT, Test of Cure, Negative | 697 | 669
  NIT, Test of Cure, Positive: number analyzed (Participants) | 719 | 727
  NIT, Test of Cure, Positive | 22 | 58
  LEU, Baseline, Negative: number analyzed (Participants) | 789 | 782
  LEU, Baseline, Negative | 245 | 232
  LEU, Baseline, Trace: number analyzed (Participants) | 789 | 782
  LEU, Baseline, Trace | 96 | 91
  LEU, Baseline, Small: number analyzed (Participants) | 789 | 782
  LEU, Baseline, Small | 75 | 80
  LEU, Baseline, Moderate: number analyzed (Participants) | 789 | 782
  LEU, Baseline, Moderate | 120 | 116
  LEU, Baseline, Large: number analyzed (Participants) | 789 | 782
  LEU, Baseline, Large | 251 | 262
  LEU, Baseline, Missing: number analyzed (Participants) | 789 | 782
  LEU, Baseline, Missing | 2 | 1
  LEU, On-Therapy, Negative: number analyzed (Participants) | 731 | 737
  LEU, On-Therapy, Negative | 510 | 475
  LEU, On-Therapy, Trace: number analyzed (Participants) | 731 | 737
  LEU, On-Therapy, Trace | 79 | 82
  LEU, On-Therapy, Small: number analyzed (Participants) | 731 | 737
  LEU, On-Therapy, Small | 50 | 49
  LEU, On-Therapy, Moderate: number analyzed (Participants) | 731 | 737
  LEU, On-Therapy, Moderate | 34 | 57
  LEU, On-Therapy, Large: number analyzed (Participants) | 731 | 737
  LEU, On-Therapy, Large | 58 | 74
  LEU, Test of Cure, Negative: number analyzed (Participants) | 719 | 727
  LEU, Test of Cure, Negative | 526 | 494
  LEU, Test of Cure, Trace: number analyzed (Participants) | 719 | 727
  LEU, Test of Cure, Trace | 61 | 49
  LEU, Test of Cure, Small: number analyzed (Participants) | 719 | 727
  LEU, Test of Cure, Small | 43 | 48
  LEU, Test of Cure, Moderate: number analyzed (Participants) | 719 | 727
  LEU, Test of Cure, Moderate | 35 | 59
  LEU, Test of Cure, Large: number analyzed (Participants) | 719 | 727
  LEU, Test of Cure, Large | 54 | 77

29. Secondary Outcome: Absolute Mean Values of Urine Specific Gravity
Description: Urine samples were collected from participants to assess urine specific gravity. Baseline is defined as the latest pre-dose assessment with a non-missing value.
Time Frame: Baseline (on or before Day 1), On-Therapy (Days 2 to 5), and Test of cure (Days 9 to 16)
Population: Safety population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Gepotidacin | Nitrofurantoin
Number analyzed (Participants) | 779 | 773
Ratio
  Baseline | 1.0172 (0.00693) | 1.0174 (0.00686)
  On-Therapy: number analyzed (Participants) | 731 | 737
  On-Therapy | 1.0176 (0.00716) | 1.0167 (0.00696)
  Test of Cure: number analyzed (Participants) | 719 | 727
  Test of Cure | 1.0179 (0.00712) | 1.0179 (0.00719)

30. Secondary Outcome: Absolute Mean Values of Urine Potential of Hydrogen (pH)
Description: Urine samples were collected from participants to assess urine pH levels. Baseline is defined as the latest pre-dose assessment with a non-missing value.
Time Frame: Baseline (on or before Day 1), On-Therapy (Days 2 to 5), and Test of cure (Days 9 to 16)
Population: Safety population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: pH
Arm/Group | Gepotidacin | Nitrofurantoin
Number analyzed (Participants) | 763 | 764
pH
  pH, Baseline | 5.7 (0.8) | 5.7 (0.79)
  pH, On-Therapy: number analyzed (Participants) | 726 | 733
  pH, On-Therapy | 5.6 (0.66) | 5.6 (0.69)
  pH, Test of Cure: number analyzed (Participants) | 716 | 726
  pH, Test of Cure | 5.6 (0.69) | 5.7 (0.71)

31. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) at On-Therapy and Test of Cure Visit
Description: SBP and DBP were measured in a semi-supine position after 5 minutes rest. Baseline is defined as the latest pre-dose assessment with a non-missing value.
Time Frame: Baseline (on or before Day 1), On-Therapy (Days 2 to 5), and Test of cure (Days 9 to 16)
Population: Safety population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Gepotidacin | Nitrofurantoin
Number analyzed (Participants) | 804 | 798
Millimeters of mercury (mmHg)
  SBP, Baseline | 122 (13.33) | 122.7 (13.98)
  SBP, On-Therapy: number analyzed (Participants) | 745 | 751
  SBP, On-Therapy | -1.1 (10.14) | -1.1 (10.72)
  SBP, Test of Cure: number analyzed (Participants) | 732 | 752
  SBP, Test of Cure | -0.4 (11.67) | -1.8 (12.19)
  DBP, Baseline | 76.9 (8.17) | 77 (9)
  DBP, On-Therapy: number analyzed (Participants) | 745 | 751
  DBP, On-Therapy | -0.5 (7.30) | -0.6 (7.73)
  DBP, Test of Cure: number analyzed (Participants) | 732 | 752
  DBP, Test of Cure | -0.1 (7.98) | -1.3 (8.37)

32. Secondary Outcome: Change From Baseline in Pulse Rate at On Therapy and Test of Cure Visit
Description: Pulse rate was measured in a semi-supine position after 5 minutes rest. Baseline is defined as the latest pre-dose assessment with a non-missing value.
Time Frame: Baseline (on or before Day 1), On-Therapy (Days 2 to 5), and Test of cure (Days 9 to 16)
Population: Safety population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | Gepotidacin | Nitrofurantoin
Number analyzed (Participants) | 804 | 798
beats per minute (bpm)
  Pulse rate, Baseline | 73.2 (9.64) | 73.7 (10.32)
  Pulse rate, On-Therapy: number analyzed (Participants) | 745 | 751
  Pulse rate, On-Therapy | 0.9 (8.24) | 1.3 (8.66)
  Pulse rate, Test of Cure: number analyzed (Participants) | 732 | 752
  Pulse rate, Test of Cure | 1.8 (9.74) | 1.7 (9.95)

33. Secondary Outcome: Change From Baseline in Body Temperature
Description: Temperature was measured in a semi-supine position after 5 minutes rest. Baseline is defined as the latest pre-dose assessment with a non-missing value.
Time Frame: Baseline (on or before Day 1), On-Therapy (Days 2 to 5), and Test of cure (Days 9 to 16)
Population: Safety population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Celsius
Arm/Group | Gepotidacin | Nitrofurantoin
Number analyzed (Participants) | 804 | 798
Celsius
  Temperature, Baseline | 36.61 (0.346) | 36.63 (0.317)
  Temperature, On-Therapy: number analyzed (Participants) | 744 | 751
  Temperature, On-Therapy | -0.01 (0.334) | -0.01 (0.372)
  Temperature, Test of Cure: number analyzed (Participants) | 732 | 752
  Temperature, Test of Cure | -0.01 (0.349) | -0.04 (0.351)

34. Secondary Outcome: Number of Participants With Maximum Change From Baseline in Electrocardiograms (ECG) Parameter: QT Interval Corrected for Heart Rate According to Bazett's Formula (QTcB) at Worst-case Post-baseline
Description: Triplicate 12-lead ECGs (over an approximate 5- to 10-minute period) were performed using an ECG machine. Baseline is defined as the latest pre-dose assessment with a non-missing value. The row titles <=450, >450 to <=480, >480 to <=500 millisecond (msec) are the values at baseline. The category titles <= 30, 31-60, >60 msec are the maximum change from baseline values. The maximum change from baseline value category was determined by comparing the baseline value category to the worst-case post-baseline value category for each participant, which considered unscheduled and out of visit window assessments. Data of number of participants with any change at worst-case post-baseline (maximum grade increase post-baseline) is presented.
Time Frame: Up to Day 31
Population: Safety population. Only those participants with data available at the specified data points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Gepotidacin | Nitrofurantoin
Number analyzed (Participants) | 791 | 784
Participants
  <= 450 msec: number analyzed (Participants) | 746 | 743
  <= 450 msec: <=30 msec | 675 | 700
  <= 450 msec: 31-60 msec | 23 | 12
  <= 450 msec: >60 msec | 1 | 0
  <= 450 msec: Missing | 47 | 31
  >450 to <=480 msec: number analyzed (Participants) | 45 | 40
  >450 to <=480 msec: <=30 msec | 40 | 37
  >450 to <=480 msec: 31-60 msec | 2 | 0
  >450 to <=480 msec: >60 msec | 0 | 0
  >450 to <=480 msec: Missing | 3 | 3
  >480 to <=500 msec: number analyzed (Participants) | 0 | 1
  >480 to <=500 msec: <=30 msec |  | 1
  >480 to <=500 msec: 31-60 msec |  | 0
  >480 to <=500 msec: >60 msec |  | 0
  >480 to <=500 msec: Missing |  | 0

35. Secondary Outcome: Number of Participants With Maximum Change From Baseline in Electrocardiograms (ECG) Parameter- QT Interval Corrected for Heart Rate According to Fridericia's Formula (QTcF) at Worst-case Post-baseline
Description: Triplicate 12-lead ECGs (over an approximate 5- to 10-minute period) were performed using an ECG machine. Baseline is defined as the latest pre-dose assessment with a non-missing value. The row titles <=450 msec, >450 msec to <=480 msec are the values at baseline. The category titles <= 30, 31-60, >60 msec are the maximum change from baseline values. The maximum change from baseline value category was determined by comparing the baseline value category to the worst-case post-baseline value category for each participant, which considered unscheduled and out of visit window assessments. Data of number of participants with any change at worst-case post-baseline (maximum grade increase post-baseline) is presented.
Time Frame: Up to Day 31
Population: Safety population. Only those participants with data available at the specified data points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Gepotidacin | Nitrofurantoin
Number analyzed (Participants) | 791 | 784
Participants
  <= 450 msec: number analyzed (Participants) | 783 | 779
  <= 450 msec: <=30 msec | 721 | 742
  <= 450 msec: 31-60 msec | 12 | 4
  <= 450 msec: >60 msec | 0 | 0
  <= 450 msec: Missing | 50 | 33
  >450 to <=480 msec: number analyzed (Participants) | 8 | 5
  >450 to <=480 msec: <=30 msec | 8 | 4
  >450 to <=480 msec: 31-60 msec | 0 | 0
  >450 to <=480 msec: >60 msec | 0 | 0
  >450 to <=480 msec: Missing | 0 | 1

ADVERSE EVENTS:
Time Frame: All cause mortality, non-serious adverse events (Non-SAEs) and serious adverse events (SAEs) were collected from the time of first dose (Day 1) through the final follow-up visit (Day 21-31)
Description: Safety population included all randomized participants who receive at least 1 dose of study treatment.
Arm/Group | Gepotidacin | Nitrofurantoin
All-Cause Mortality (participants affected / at risk) | 0/804 | 0/798
Serious Adverse Events (participants affected / at risk) | 5/804 | 5/798
Other Adverse Events (participants affected / at risk) | 235/804 | 119/798
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gepotidacin (N=804) | Nitrofurantoin (N=798)
Atrial fribrillation (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 2 (2) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 2 (2)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gepotidacin (N=804) | Nitrofurantoin (N=798)
Diarrhoea (Gastrointestinal disorders) | 147 (166) | 24 (25)
Nausea (Gastrointestinal disorders) | 65 (66) | 35 (36)
Flatulence (Gastrointestinal disorders) | 28 (29) | 4 (4)
Faeces soft (Gastrointestinal disorders) | 23 (30) | 4 (4)
Vomiting (Gastrointestinal disorders) | 18 (18) | 7 (7)
Abdominal pain (Gastrointestinal disorders) | 12 (12) | 7 (8)
Abdominal discomfort (Gastrointestinal disorders) | 9 (9) | 4 (5)
Headache (Nervous system disorders) | 21 (23) | 22 (27)
Dizziness (Nervous system disorders) | 18 (18) | 11 (12)
Urinary tract infection (Infections and infestations) | 11 (11) | 15 (15)
Fungal infection (Infections and infestations) | 9 (9) | 10 (10)
COVID-19 (Infections and infestations) | 9 (9) | 5 (6)
Fatigue (General disorders) | 3 (3) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-11-03): https://cdn.clinicaltrials.gov/large-docs/44/NCT04187144/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-14): https://cdn.clinicaltrials.gov/large-docs/44/NCT04187144/SAP_001.pdf